CLINICAL TRIAL: NCT05160610
Title: Improving Thrombolysis Implementation Based on Electronic Monitoring in Acute Ischemic Stroke (ITEM): a Cluster Randomized Controlled Trial
Brief Title: Improving Thrombolysis Implementation Based on Electronic Monitoring in Acute Ischemic Stroke (ITEM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITEM
Record Dates: First submitted 2021-11-16; First posted 2021-12-16 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-01

CONDITIONS: Thrombolysis Rate
Keywords: Acute ischemic stroke; Electronic monitoring; Intravenous thrombolysis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): receiving multilevel intervention, electronic monitoring and stroke registry participation
  Interventions: Behavioral: Multilevel intervention
- Control group (No Intervention): receiving routine care , electronic monitoring and stroke registry participation

INTERVENTIONS:
Behavioral: Multilevel intervention — Multilevel intervention based on AACTT theory
  Arms: Intervention group

SUMMARY:
A cluster randomized controlled trial will be conducted. Hospitals in Zhejiang Province, China, will be randomized into two arms (1:1): an intervention arm and a control arm.

Hospitals in the intervention arm will receive a multilevel intervention based on the AACTT theory, whereas hospitals in the control arm will receive no intervention and maintain routine care. All the hospitals will receive electronic monitoring. Hospitals with no stroke center or with <20 cases received thrombolysis per year will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presented with clinical signs of acute ischemic stroke within 4.5 hours of stroke onset
2. Patient's age is >18 years

Exclusion Criteria:

Contraindication for intravenous thrombolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2720 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Thrombolysis rate within 4.5 hours | Up to 4.5 hours
  The proportion of acute ischemic stroke patients within 4.5 hours of onset

SECONDARY OUTCOMES:
Thrombolysis rate within 3 hours | Up to 3 hours
  The proportion of acute ischemic stroke patients within 3 hours of onset
Excellent neurological outcomes | At 90 days
  Score of 0 to 1 on the modified Rankin Scale, on which scores range from 0 (no neurologic deficit) to 6 (death)
Favorable neurological outcomes | At 90 days
  Score of 0 to 1 on the modified Rankin Scale, on which scores range from 0 (no neurologic deficit) to 6 (death)
modified Rankin Scale score | At 90 days
  The distribution of modified Rankin Scale score at 90 days, on which scores range from 0 (no neurologic deficit) to 6 (death)
All-cause death rate | At 90 days
  All-cause death rate at 90 days
Hemorrhagic transformation | At 7 days
  the presence of hemorrhagic transformation is defined according to European Cooperative Acute Stroke Study (ECASS) II trial
Symptomatic intracranial hemorrhage | At 7 days
  Intracranial hemorrhage at 24 hours associated with an increase of ≥4 points of NIHSS score from baseline, according to European Cooperative Acute Stroke Study (ECASS) II trial
Door-to-image time | Up to 4.5 hours
  The time between hospital arrival and the initiation of image

OTHER OUTCOMES:
the proportion of acute ischemic stroke patients with Door-to-Needle Time≤60min | Up to 4.5 hours
  Difference between intervention arm and control arm in the percentage of patients receiving thrombolysis within 60 minutes of stroke onset
Door-to-needle time | Up to 4.5 hours
  The time between hospital arrival and the initiation of IVT
Onset-to-needle time | Up to 24 hours
  The time between the symptom onset and the initiation of IVT

CONTACTS AND LOCATIONS:
Overall Officials: Zexin Chen, Principal Investigator — Ethics committee the second affiliated hospital, school of medicine, Zhejiang University, China
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China